CLINICAL TRIAL: NCT04895670
Title: Empowering Youth Aging Out of Foster Care: Community Engaged Technology Solutions to Improve Transitions to Independent Living
Brief Title: Empowering Youth Aging Out of Foster Care
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Children's Health (Other)
Responsible Party: Principal Investigator, Kimberly Stone, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: 33699
Record Dates: First submitted 2021-05-01; First posted 2021-05-20 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Empowering Youth Aging out of Foster Care — App that allows storage of health information, and access to reputable health information and community resources.

SUMMARY:
Improving the health literacy of adolescents and increasing the success of transitions to adulthood from foster care are two defined Healthy People 2030 public health priorities. Skills to promote health literacy and independent living are often lacking in adolescents in foster care and young adults who have aged out of care. Frequent placement changes, no permanent home, lack of trust in adults and systems of care prevent the development of a strong support system for transitioning to adulthood from foster care, which can result in lack of access to personal health information, complicated identity documents, and disconnected child welfare, health care and community resources. These factors limit the ability to transition to adulthood successfully, drive disparities in health outcomes, and may explain lack of educational attainment and career development for young adults formerly in care. Successful transitions to independent living are unattainable unless barriers are addressed with a multidisciplinary, community-based approach.

The Rees-Jones Center for Foster Care Excellence at Children's Health and the Krissi Holman Family Resource Library at Children's Health recognized the unique needs of adolescents in foster care and young adults formerly in care (AYAFC) as they transition to independent living. We developed a partnership with community agencies (Empowering Youth Taskforce) that support these youth in the areas of child welfare (TX Department of Family and Protective Services), education (UNT PuSH Program), career development and housing support (TRAC at City Square, Zoie's Place), legal support (SMU Dedman Law School), and others, to increase AYAFC health literacy, access to health care, and awareness and use of available community resources. Frequent placement changes and unstable housing make it difficult for AYAFC to keep their health information, identity records and personal documents together, which is critical for accessing health services, enrolling in health insurance, and maintaining wellness. Since many have access to a smart phone, using technology is one way to promote adolescent health and wellness. An app is a possible solution to address many of the barriers that impede successful transition to independent living.

The goal of this project is to engage AYAFC and stakeholders who support these young people throughout North Texas to collaboratively design an app to support the transition from foster care to adulthood. This project will utilize a mixed methods approach to inform the transition process while addressing both individual and systems level barriers to increase the success of AYAFC's transition to independent living. This project builds upon work done by a multidisciplinary community task force led by the Principal Investigator, and the development of an adolescent transition process at the Rees-Jones Clinic. Community partners are fully engaged in the design of the intervention and will be involved in AYAFC and stakeholder recruitment, data analysis, and interpretation of the results.

DETAILED DESCRIPTION:
This project is uniquely community-based as the only known digital information-sharing project that will solicit input directly from AYAFC and multiple community stakeholders. Prior studies had input from youth in care, child welfare personnel and health care providers; our project includes stakeholders involved in life skills and employment training, housing support, legal advocacy, and education for a more robust community perspective. Other information sharing resources have been web-based, which is more challenging to access, or resulted in a paper guidebook. Our innovative app maximizes ease of access and portability without requiring significant cellular data usage. Assessing the health literacy skills of AYAFC can inform future interventions to support transitions to wellness in adulthood while youth are still in foster care.

This project is supported by the Region 3 Foster Care Consortium, a coalition of organizations and individuals committed to improving the lives of children involved in the foster care system. The Empowering Youth Task Force members are community partners who specialize helping youth in foster care successfully transition to adulthood. Each member organization contributes expertise on specific issues surrounding AYAFC they serve. They will engage in participant recruitment, app design and dissemination. Members of the Empowering Youth Task Force include:

The Rees-Jones Center for Foster Care Excellence is a community leader in clinical care, policy and advocacy and research. Roles include project design; development focus group questions; focus group and survey data collection and analysis; expertise on adolescent transitions from the medical provider, behavioral health provider, foster parent, and caseworker perspective; stakeholder engagement, and information dissemination.

The Krissi Holman Family Resource Library at Children's Health provide expertise in literature review and health literacy. Roles include project design; development focus group questions; survey and focus group and data collection and analysis. They will provide links to reliable health information and resources, and plain language educational materials that can be utilized through the app.

The Transition Resource Action Center at City Square supports transition-age youth with employment, education and housing, providing perspective on the issues facing young adults aging out of foster care.

The Southern Methodist University Dedman Law School Child Advocacy Clinic is a community expert on legal issues for youth aging out of foster care and will provide information resources (letter of support attached) The University of North Texas' Persevere UNTil Success Happens (PUSH) Program supports former foster youth and will provide additional perspectives on the needs of youth transitioning out of care.

The Texas Department of Family and Protective Services and their Child Protective Services and Preparation for Adult Living Program contributes expertise in child welfare transition services available to youth.

Superior Star Health Transition Services provides expertise in health insurance and support for AYAFC and will provide perspective regarding youth engagement in health insurance.

Additional community partners include Dallas Court-Appointed Special Advocates (CASA) and Zoie's Place, who provide information as unbiased child advocates and perspective about needs surrounding life skills training, support and transitional housing for AYAFC, respectively.

Study Design Most AYAFC have phones. An app is an ideal tool to help them manage reputable sources for health education and information, document storage, and access to community and child welfare resources. A community-engaged approach with AYAFC with first-hand knowledge of the foster care system will result in an app that is relevant and acceptable.

4.1 Study Design: Aim 1: Using mixed methods, (survey and focus groups) conduct a needs assessment that measures health literacy and assesses health information, supportive care, and resource needs for AYAFC transitioning from foster care to independent living.

Evaluation Methods: Survey of AYAFC to assess health literacy skills, assessment of knowledge of health and community resources, attitudes surrounding available resources and confidence in accessing digital information. Focus groups with AYAFC and community stakeholders to assess current needs surrounding health literacy, health information and community resources.

AYAFC Inclusion Criteria for all focus groups and surveys: 1) AYAFC: English-speaking, ages 18-24 who live in Texas Region 3.

Community stakeholders Inclusion Criteria (focus groups): English-speaking adults (18+) who support AYAFC (e.g. caregivers, medical, legal, and social service professionals)

Aim 2: App Development and Implementation: App development and implementation will use a user-centered design approach. This involves a needs assessment and targeted user feedback to develop an app framework. After legal approval, app infrastructure, capabilities and functionality are developed, design build-out and front and back-end integration occurs. User acceptability testing occurs at each step with testing and piloting before full roll-out.

Evaluation method: (a) Survey of implementation outcomes. (b) 4 additional focus groups with AYAFC and community stakeholders to assess attitudes toward app content, design, and usability.

Aim 3: By survey, reassess health literacy skills, and knowledge, attitudes, and confidence in accessing health information and needs for community resources.

ELIGIBILITY:
Inclusion Criteria:

* Young Adults In extended care foster care or aged out of foster care
* English-speaking
* Ages 18-24
* Community stakeholders who are English-speaking adults (18-65) who support -Adolescents and Young Adults in Foster Care or aged out of care.
* (e.g. caregivers, medical, legal, and social service professionals

Exclusion Criteria:

* Age less than 18 years old
* never in foster care.

No direct contact with Adolescents and Young Adults in Foster Care or aged out of care.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 40% of adolescents in foster care have a chronic health problem or significant mental health diagnosis; many take medications daily. One third of adolescents in foster care do not have a permanent home prior to turning 18. They often have multiple placement changes, extended involvement in the child welfare system and substantial neglect, abuse and trauma histories. They may lack trust in adults, systems of care and ongoing support as they transition to adulthood. They also may lack access to their health information, identity documents and resources needed to successfully transition to adulthood. In 2019, over 1,100 children aged out of care in Texas. Almost 25% of children aging out of foster care had been in care before they were teenagers; many were in group homes or shelters and had multiple foster care placements. In Texas, youth who aged out of foster care are less likely to finish high school, go to college or be employed than youth not in care.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Needs assessment for app development | 24 months
  Qualitatively assess by focus group needs and features for app to assist in management of health information and access of health information and community resources.
Impact of app use on Health Literacy | 12 months
  Measured by pre and post health literacy assessment.
Impact of app use on Knowledge of Health Information and Community Resources | 6 months
  Measured by pre and post knowledge assessment
App Acceptability | 6 months
  Qualitative Data Collection by Focus Group regarding app usability and acceptability.
App Engagement | 6 months
  Measured by number of app usages.
App Use | 6 months
  Measured by time spent accessing data

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens Health, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No